CLINICAL TRIAL: NCT03159572
Title: Homologous Recombination Inquiry Through Ovarian Malignancy Investigations
Acronym: HITOMI
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Department of Obstetrics and Gynecology, School of Medicine, Niigata University (Unknown); Japanese Gynecologic Oncology Group (Other); Tohoku Medical Megabank Organization(ToMMo) (Unknown)
Responsible Party: Sponsor
Other Study IDs: JGOG3025; UMIN000026303 (Other: UMIN-CTR)
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Ovarian cancer; Fallopian tube cancer; Primary peritoneal cancer; Germline Breast Cancer Susceptibility Gene (BRCA1/2 gene); Homologous Recombination Deficiency (HRD)
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ovarian cancer group: Patients who are diagnosed with ovarian cancer and have a plan of surgery.

SUMMARY:
To investigate the frequency and clinical significance of Homologous Recombination Deficiency (HRD) in Japanese patients with ovarian cancer (including Fallopian tube cancer and primary peritoneal cancer).

DETAILED DESCRIPTION:
In this study, investigators plan to clarify the frequency of Homologous Recombination Deficiency (HRD) in Japanese patients with ovarian cancer (including fallopian tube cancer and primary peritoneal cancer).

And investigators will also investigate whether HRD-positive ovarian cancer patients show the clinical characteristics of highly platinum-sensitivity and good prognosis, comparing to HRD-negative ovarian cancer patients.

In addition, it is planned to investigate any association between Progression Free Survival (PFS) / Platinum-Sensitivity and germline mutation in Breast Cancer Susceptibility Gene (BRCA1/2 gene) in ovarian cancer patients who can provide the patients' gBRCA1/2 gene information for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who can approve informed consent and sign it. Patients who show their will to participate in this study and can sign the informed consent forms by themselves.
2. Patients who are clinically diagnosed as having ovarian cancer and can provide written informed consent before the surgery.
3. Patients who can provide tumor tissue specimens. (except ascites cytology and cell block specimens)
4. Patients who are 20 years old and over at the enrollment.
5. Patients with ECOG Performance status (PS): 0-2.

Exclusion Criteria:

1. Patients with active concomitant malignancy* except breast cancer.

   *Includes synchronous multiple cancer and metachronous multiple cancer with less than 5 years of disease free survival. However, excludes skin basal cell carcinoma, skin squamous cell carcinoma, and any other curable lesions with local therapy such as carcinoma in situ or intramucosal carcinoma.
2. Patients who are diagnosed as any other acute/chronic, physically/mentally severe diseases and judged by the primary physician as inappropriate to enroll this study because of safety reasons or any influence to study outcomes.
3. Any other cases that are inappropriate to enroll this study, judged by study principal investigator.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ovarian cancer patients who provided written informed consent including providing tumor tissue specimens before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 996 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Frequency of HRD in patients with ovarian cancer (including fallopian tube cancer and primary peritoneal cancer) | 17 months
  When all tumor samples are stored at ToMMo after the term of registration, DNA are extracted from frozen tumor tissue. These extracted tumor DNA, after confirmed at inspection body that it has constant qualities, are examined for HRD by DNA target sequencing.

SECONDARY OUTCOMES:
Association between Progression Free Survival (PFS) / Response Rate and HRD in patients with ovarian cancer (including fallopian tube cancer and primary peritoneal cancer) | 48 months
  PFS is calculated from registration date to the date diagnosed as progression or the date of death from any cause, whichever comes earlier. Response rate(RR) is determined the rate of patients who are evaluated of best overall response as CR(complete response) or PR(partial response) from those with measurable disease (based on Guidelines to Evaluate the Response to Treatment in Solid Tumors, RESIST).
  Association between PFS/RR and HRD which is clarified as primary outcome is assessed.
Association between Progression Free Survival (PFS) / Response Rate and germline mutation in BRCA1/2 gene in patients with ovarian cancer (including fallopian tube cancer and primary peritoneal cancer) | 48 months
  PFS is calculated from registration date diagnosed as having progression or the date of death from any cause, whichever comes earlier. Response rate(RR) is determined the rate of patients who are evaluated of best overall response as CR(complete response) or PR(partial response) from those with measurable disease (based on Guidelines to Evaluate the Response to Treatment in Solid Tumors, RESIST).
  Association between PFS/RR and gBRCA1/2 gene information from patients who can provide their gBCRA1/2 gene information with their informed consent, is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Enomoto, MD, Ph.D, Study Chair — Department of Obstetrics and Gynecology, Niigata University Graduate School of Medical and Dental Sciences
Locations (1):
- Niigata University Graduate School of Medical and Dental Sciences, Niigata, Niigata, Japan

IPD SHARING:
Plan to Share IPD: Undecided